CLINICAL TRIAL: NCT03210597
Title: Effects of Water-Based Aerobic Training, Resistance Training and Concurrent Training in Women With Metabolic Syndrome: A Randomized Controlled Trial
Brief Title: Effects of Water-Based Exercise in Women With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Luiz Fernando Martins Kruel, Doctor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP UFRGS 1.499.603
Record Dates: First submitted 2017-06-22; First posted 2017-07-07 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Metabolic Syndrome
Keywords: water-base exercise
MeSH Terms: conditions — Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant: During the training period the subjects were not informed about the training modality they were performing and also were not informed about the modalities of the other subjects, only they were informed that hydrogymnastic sessions would be performed.
  Outcomes assessor:The team evaluating the outcomes was blinded, not receiving information about the intervention received by the subjects participating in the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hydro-aerobic (Experimental): Water aerobics exercise
  Interventions: Other: Exercise
- hydro-power (Experimental): Resistance water exercise
  Interventions: Other: Exercise
- hydro-combined (Experimental): Water aerobics and resistance water exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The subjects performed training in aquatic environment

SUMMARY:
The objective of the present study was to compare the neuromuscular, cardiorespiratory and metabolic effects of 12 weeks of aerobic training, strength training and combined training in the aquatic environment in women with MS. For this purpose, 51 postmenopausal, sedentary and MS women were randomly divided into three intervention groups: hydro-aerobic (HA, n = 18, 63.77 ± 5.03 years), hydro-power (HF, n = 16, 61.01 ± 4.93 years) and hydro-combined (HC; n = 17; 60.52 ± 6.91). A subsample participated in eight weeks without physical exercise to characterize a control period. The three intervention groups performed two weekly sessions of 60 minutes for 12 weeks. Before and after the training period, blood tests, muscle strength tests, cardiorespiratory evaluation, functional tests and a questionnaire were performed. For statistical analysis, the Generalized Estimates Equations (GEE) model was used, using the "group" and the "time" as factors. The Bonferroni post hoc was used to locate the differences and the significance index adopted was α = 0.05.

DETAILED DESCRIPTION:
Water-based exercise as a mode of aquatic exercise has been highlighted in the scientific literature. Research on different models of training, aerobic, muscle strength and combined (aerobic and muscle strength), have already demonstrated their beneficial effects on different physical abilities. Recent studies indicate benefits of water-based exercise for the population with metabolic diseases such as hypertension, type 2 diabetes, dyslipidemias and obesity. However, for subjects with metabolic syndrome (MS) there are few studies that investigated which training model in the aquatic environment could generate physical and metabolic improvements.

This study is characterized as a randomized clinical trial, which treated three intervention groups with physical exercise programs. A subsample participated in a period of eight weeks without physical exercise to characterize a control period. The subjects in this subsample were later randomized into the intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal;
* Sedentary;
* Presented at least three positive components within the five possible to characterize the metabolic syndrome.

Exclusion Criteria:

* Smokers.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure | 12 weeks
  mmHg

SECONDARY OUTCOMES:
Strength tests: Maximum dynamic muscle strength | 12 weeks
  One repetition test: how many kilograms the subject is able to withstand on a repetition of elbow flexion and knee extension exercise
EMG test | 12 weeks
  Maximum isometric amplitude of the electromyographic signal of the vastus lateralis and rectus femoris muscles
Time Up and go test | 12 weeks
  How long (in seconds) the subject needs to lift from a chair, walk 2.44 meters, and sit in a chair again
Sit and Stand test | 12 weeks
  How often in 30 seconds the subject is able to get up and sit on a chair.
Triglyceride levels | 12 weeks
  blood test: mg/dl
HDL cholesterol levels | 12 weeks
  blood test: mg/dl
Fasting blood glucose levels | 12 weeks
  blood test: mg/dl
Waist circumference | 12 weeks
  centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Luiz F. Martins Kruel, Study Director — Federal Universty of Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No